CLINICAL TRIAL: NCT00641589
Title: An Open-Label, Randomized Study to Determine the Pharmacokinetic and Pharmacodynamic Profiles of PROCRIT (Epoetin Alfa) in Anemic Subjects With Chronic Kidney Disease
Brief Title: A Study to Determine the Pharmacokinetic and Pharmacodynamic Profiles of PROCRIT (Epoetin Alfa) in Anemic Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Centocor Ortho Biotech Services, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002299
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Kidney Disease; Anemia
Keywords: Chronic Kidney Disease; anemia; epoetin alfa
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The primary objective of this study is to describe how four different dosing regimens of PROCRIT (epoetin alfa) are utilized in patients with anemia due to non-dialysis chronic kidney disease (CKD).

DETAILED DESCRIPTION:
This is a prospective, open-label (both the patient and the physician know the drug and drug dose being given), randomized (patients are assigned to a dosing regimen by chance), multicenter, pharmacokinetic study in patients with anemia secondary to non-dialysis chronic kidney disease (CKD). A pharmacokinetic study is one that evaluates the process by which a drug is utilized by the body.

Approximately 40 patients will participate in this study. This study has 3 Phases; the Screening Phase, the Open-Label Treatment Phase and Study Completion/Early Withdrawal Phase. In the Screening Phase, patients may be evaluated up to 14 days before study entry. The Treatment Phase begins when the patient is randomly assigned to a treatment group and continues until the patient has received the last dose of study drug. The Study Completion/Early Withdrawal Phase is the phase during which the last study-related procedures take place. This Phase should occur on Study Day 64 for the Q4W group and on Study Day 36 for all other dosing regimens. Patients who satisfy all study inclusion and exclusion criteria and consent to participate in the study will be randomly assigned to one of four treatment groups. Dosing will continue through Study Day 26 for treatment group A, through Study Day 22 for treatment group B, through Study Day 15 for treatment group C, and through Study Day 29 for treatment group D. No dose escalation or dose reductions are allowed during the study. Safety will be monitored by physical examinations, vital signs, clinical laboratory tests, and the occurrence and severity of any adverse events. Safety monitoring will continue through 30 days after the last visit for all treatment groups.

Pharmacokinetic and pharmacodynamic (the study of the action or effects of drugs on the body) sampling will occur throughout the study. A patient evaluable for pharmacokinetic and pharmacodynamic parameters is one who receives the first scheduled dose of the assigned study drug, has at least 75% of the pharmacokinetic samples collected up to and including Day 29 for all groups, and does not receive any red blood cell (RBC) transfusions prior to Study Day 8. Pharmacokinetic evaluations will continue through Study Day 29 for groups A, B, C; through Study Day 57 for Group D, and will include but are not limited to: maximal serum concentrations of erythropoietin, time to reach maximal serum concentration and time for erythropoietin to be eliminated from the body. Pharmacodynamic evaluations continue through Study Day 36 for Groups A,B,C; through Study Day 64 for Group D, and will include but are not limited to hemoglobin (Hg), hematocrit (Hct), total red blood cell (RBC) count. The primary objective of this study is to describe the pharmacokinetic profiles of four different dosing regimens of PROCRIT (epoetin alfa) in patients with anemia secondary to non-dialysis chronic kidney disease (CKD).

The secondary objective is to describe the pharmacodynamic response to the four epoetin alfa study dosing regimens. Patients will be randomly assigned to one of four dosing regimens of epoetin alfa: Group A: 50 IU (International Units)/kilogram (kg) three times per week (TIW); Group B: 10,000 IU once weekly (QW); Group C: 20,000 IU every 2 weeks (Q2W); and Group D: 40,000 IU every 4 weeks (Q4W).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Glomerular Filtration Rate (GFR) within 15-60 mL/min/1.73m2 and stable creatinine over the past 6 months and no expected need for dialysis during the study
* Patients with a hemoglobin (Hg) < 11 g/dL at Screening
* Patients with a transferrin saturation >= 20% or a ferritin >= 50 ng/mL.
* Patients who have not received any erythropoietic agents within 6 weeks prior to the first study dose
* Patients with reproductive potential must have a negative B-HCG pregnancy test within 14 days of the first dose of study drug and a negative urine pregnancy test on the day of the first dose of study drug
* Patients and their partners must be practicing an effective method of birth control before entry and throughout the study

Exclusion Criteria:

* Exclusion criteria include but are not limited to the following: Patients with significant hematological disease (disorders of the blood and blood forming tissues
* including but not limited to myelodysplastic syndrome, hematological malignancy, hemolytic syndromes, hemoglobinopathy)
* Patients with liver function test results > 2 or more times the normal value
* Patients with new onset seizures (within the last 3 months) or seizures not controlled by medication prior to admission in to the study
* Patients with a history of thrombotic vascular events (including by not limited to acute myocardial infarction (AMI) within the previous 6 months, stroke, transient ischemic attack (TIA), deep vein thrombosis,(DT) and pulmonary embolism (PE)
* Patients with poorly controlled or uncontrolled hypertension
* Patients with anemia due to blood loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to describe the pharmacokinetic (PK) profiles of 4 different dosing regimens of PROCRIT in patients with anemia secondary to chronic kidney disease (CKD) not on dialysis.

SECONDARY OUTCOMES:
The secondary objective is to describe the pharmacodynamic (PD) response to the four PROCRIT study dosing regimens using the following outcomes: absolute and % reticulocyte count, hemoglobin (Hb), hematocrit (Hct), and red blood cell (RBC) count.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An open-label, randomized study to deteremine the pharmacokinetic and pharmacodynamic profiles of PROCRIT (Epoetin alfa) in anemic subjects with chronic kidney disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=468&filename=CR002299_CSR.pdf